CLINICAL TRIAL: NCT03578861
Title: Development and Pilot Testing of a Dementia Specific Respite Care Concept With Scope on Mobility and Couseling.
Brief Title: Dementia Specific Respite Care Concept.
Acronym: DESKK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WI025
Record Dates: First submitted 2018-06-18; First posted 2018-07-06 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-06

CONDITIONS: Mobility; Dementia; Counseling; Respite Care
MeSH Terms: conditions — Dementia | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia related mobility and counseling (Experimental): The DESKK mobility program is based on the already existing day structure of the RC facility with two slots a day for physical activation activities (1 ½ hours forenoon and 1 ½ hours afternoon). The program structures these activities based on specific developed exercises, which are focused on the individual mobility level of every PwD and his/her mobility level.
  The DESKK counseling program is an effort to structure and systemize counseling processes focused on the respite care setting by different documents and assessments.
  Interventions: Other: Dementia related mobility and counseling

INTERVENTIONS:
Other: Dementia related mobility and counseling — The DESKK mobility program is based on the already existing day structure of the RC facility with two slots a day for physical activation activities (1 ½ hours forenoon and 1 ½ hours afternoon). The program structures these activities based on specific developed exercises, which are focused on the individual mobility level of every PwD and his/her mobility level.
  The DESKK counseling program is an effort to structure and systemize counseling processes focused on the respite care setting by different documents and assessments.

SUMMARY:
Objectives:

Specific mobility programs can delay the functional decline in people with dementia (PwD) and help to preserve their abilities of daily living. Respite care is a common used short time inpatient service (max. 4 weeks of stay) to support dementia care arrangements. Within the DESKK project, a concept is developed which complements and optimizes dementia-specific respite care through a mobility program and a counseling program. As one part of the DESKK study, it is the aim to develop and implement a time effective and evidence based mobility program for PwD in respite care which can be individually adapted on PwD needs and preferences. It includes a short "homework-program" for caring relatives to facilitate ongoing mobility training of the PwD after returned back home.

Methods:

A pilot based, quasi-experimental evaluation study is conducted in a specialized respite care facility for PwD. The concept was developed on the basis of a comprehensive literature research, study visits at existing counseling programs as well as expert workshops with practitioners and scientists. To evaluate the implementation process, qualitative data are collected by single und group interviews. Quantitative data are collected using validated instruments to assess mobility and cognitive function of PwD. A mixed methods triangulation approach will be used to aggregate qualitative and quantitative data.

Discussion:

It is expected that the RC concept will be suitable and understandable for the staff, so that it can be implemented in the RC facility. As a result of the mobility program, the physical abilities of the PwDs should improve. Similar, the burden of the caregivers should be reduced by combined effects of the counselling program and the higher mobility level of the PwD. The whole DESKK concept, including a systematic counseling program for caring relatives, which is not part of this presentation, will be described in form of a practice friendly website to get disseminated into clinical routine after its successful evaluation.

DETAILED DESCRIPTION:
Around the world, caring relatives play the most important role in care of people with dementia (PwD) at home. In 2012 approximately 24.3 million people were affected by dementia worldwide and more than 1.5 million people are suffering from dementia in Germany. These numbers are expected to rise up significantly within the next 20 years. As a direct consequence of dementia-specific care, caring relatives are often heavily burdened. Some common symptoms of dementia include progressive and frequent memory loss as well as confusion, personality change and apathy. Furthermore, the abilities for walking and standing activities get weaker especially because of balance dysfunctions. These symptoms lead to a loss of ability to perform everyday tasks for the PwD and an increased risk of falling. Among others, this situation can destruct the stability of care arrangement at home and lead to a transfer of the PwD to long term care but most PwD have the wish to stay at home if possible.

Respite care (RC) is a common used short term inpatient service with the primary aim to support home care arrangements for PwD and their caring relatives. To reach this aim, caring relatives can bring their cared persons to a specialized RC care facility, where they can stay about 1 to 8 weeks. During this time, RC facilities could develop and implement individual tailored support interventions focused on the concerned PwD and caring relatives to reach a stabilization of their caring situation at home.

However, there are no evaluated or standardized programs for the support of PwD and caring relatives in the RC setting till today. In particular, this is a serious problem because there is an increasing number of RC residents who suffer from cognitive impairments or dementia.

An individual tailored, specific RC concept for people with dementia and their caring relatives could focus on their special needs and help to stabilize the caring situation effectively.

In an actual Cochrane review it was pointed out that there is a high demand for mobility based rehabilitation programs for PwD with significant positive effects related to mobility based ADL abilities. Mobility based interventions generate the highest effects of all other interventions, including medication, related to ADL abilities of PwD and with respect to their level of independence in general. However, few standardized and detailed described programs for mobility based interventions focused on PwD exist until today. There are no structured mobility based rehabilitation programs to support PwD and caring relatives in the RC setting. Another Cochrane review pointed out that situation does not only apply for Germany but even in international context. With scope to caring relatives, professional dementia-specific counseling services have positive effects on the psychological and psychosomatic symptoms, coping with stress and managing behavioral disturbances. To date, there is no dementia-specific counseling programs specialized to the RC setting, though RC facilities have the chance to reach caring relatives, which are often no more accessible for other dementia support services, because of their overburdened situation and thereby very little time resources. However, especially these caring relatives have a strong need for information about dementia and related support services.

Primary aim of the DESKK Study is the development, test and evaluation of a dementia specific RC concept with scope on mobility (PwD) and counseling (caring relatives) referred to its usability and implementation requirements. Furthermore an explorative outcome evaluation will be performed to describe intervention processes of this dementia specific concept focused on RC staff, PwD and caring relatives. To reach these study aims, following research questions are intended to be answered:

1. What kind of intervention parts and RC structures/processes are relevant for the development of a dementia specific RC concept focused on an ADL based mobility program for PwD and a counseling program for caring relatives?
2. How can the DESKK mobility and counseling program be developed and implemented suitable for the respite care setting?
3. What changes occur during the DESKK mobility and counseling intervention related to the PwD and caring relatives?
4. How is the DESKK concept subjective rated by the caring relatives and what changes related to burden (CR) and mobility (PwD) occurred after ending the RC stay (Follow-Up).

ELIGIBILITY:
Inclusion Criteria:

Caring relatives:

* Willingness to take part at the counseling intervention (informed consent)
* Sufficient language skills to understand the counseling sessions
* CR has to be the primary care person for the PwD

People with dementia

* Willingness to take part at the rehabilitation intervention (informed consent [if necessary: signing by the primary care person])
* Capability to understand and follow (training) instructions with support of the involved training assessors (subjective pre-assessment by raters)
* Capability to stand and walk short distances (min. 3 Meter) with support of the involved training assessors
* Minimum amount of 13 days stay in the RC center (planned)

Exclusion Criteria:

* Other severe cognitive impairments or other severe neurological disease

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | 10 min
  The SPPB can be used for the analyses of ADL related capabilities of old people related to gait performance and strength as well related to static balance. This test can also be used for people with cognitive retardation. Furthermore the Instrument is validated and reliable.

SECONDARY OUTCOMES:
Nurses' Observation Scale for Geriatric Patients (NOSGER) | 10 min
  The NOSGER Assessment is a validated and fast usable Instrument for the measurement of challenging behavior during the last 14 days. It can be filled out by nursing staff as well as by caring relatives and has an ADL focus.
Nurses' Observation Scale for Geriatric Patients (MMST) | 25 min
  The MMST is a common and validated instrument to get information about the cognitive status of persons including a rating scale which rated between not and severely cognitive impaired.
Box and Blocks Test (BBT) | 5 min
  The BBT can be used for the analyses of rough coordination skills related to the upper extremity, arms and hand. It is easy and fast to use, validated and reliable.
Strength-Dexterity Test (SD) | 2 min
  The SD is a Hand muscle strength test and can be performed very fast and easily.
Nine-Hole Peg Test (NHPT) | 2 min
  The NHPT can be used for the analyses of fine coordination relates to hands and fingers. It is easy and fast to use, validated and reliable.
Berliner Inventar zu Angehörigenbelastung-Demenz (BIZA-D) | 15 min
  The BIZA-D can be filled out relative time effective and it measures the subjective and objective burden of caring relatives of PwD. It is validated and also mobility based ADL related.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Holle, Dr, Principal Investigator — DZNE Witten
Locations (1):
- DZNE, Witten, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be available based on the informed consent of the participants. Data from the study can be requested from the first author via steffen.heinrich@dzne.de
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available in April 2019.
Access Criteria: E-Mail request via: steffen.heinrich@dzne.de
URL: https://www.dzne.de/forschung/studien/projekte-der-versorgungsforschung/deskk/

REFERENCES:
- [Background] Dassen, T. (2009). Bundesweite Erhebung zu Pflegeproblemen 2009. Studie aus Pflegeheimen und Krankenhäusern. Berlin: Charité.
- [Background] DAlzG. (2016). Informationblatt 1 - Die Häufigkeit von Demenzerkrankungen. Retrieved from https://www.deutsche-alzheimer.de/fileadmin/alz/pdf/factsheets/infoblatt1_haeufigkeit_demenzerkrankungen_dalzg.pdf
- [Background] WHO. (2012). Dementia - A public health priority. Retrieved from http://whqlibdoc.who.int/publications/2012/9789241564458_eng.pdf
- [Background] Radenbach K, Retzlik J, Meyer-Rotz SH, Wolff-Menzler C, Wolff J, Esselmann H, Godemann F, Riemenschneider M, Wiltfang J, Jessen F. [Guideline-adherent inpatient psychiatric psychotherapeutic treatment of behavioral and psychological symptoms of dementia : Normative definition of personnel requirements]. Nervenarzt. 2017 Sep;88(9):1010-1019. doi: 10.1007/s00115-016-0195-9. German. PMID 27581115
- [Background] Reggentin H. [Caregiver's burden of caring for patients with dementia in group living compared to to domestic and inpatient care]. Z Gerontol Geriatr. 2005 Apr;38(2):101-7. doi: 10.1007/s00391-005-0295-9. German. PMID 15868348
- [Background] Shea, T. (2012). Dementia - Understanding brain diseases and disorders. New York: Rosen Publishing.
- [Background] van Doorn C, Gruber-Baldini AL, Zimmerman S, Hebel JR, Port CL, Baumgarten M, Quinn CC, Taler G, May C, Magaziner J; Epidemiology of Dementia in Nursing Homes Research Group. Dementia as a risk factor for falls and fall injuries among nursing home residents. J Am Geriatr Soc. 2003 Sep;51(9):1213-8. doi: 10.1046/j.1532-5415.2003.51404.x. PMID 12919232
- [Background] Forbes D, Forbes SC, Blake CM, Thiessen EJ, Forbes S. Exercise programs for people with dementia. Cochrane Database Syst Rev. 2015 Apr 15;2015(4):CD006489. doi: 10.1002/14651858.CD006489.pub4. PMID 25874613
- [Background] Maayan N, Soares-Weiser K, Lee H. Respite care for people with dementia and their carers. Cochrane Database Syst Rev. 2014 Jan 16;2014(1):CD004396. doi: 10.1002/14651858.CD004396.pub3. PMID 24435941
- [Background] Kurz A, Hallauer J, Jansen S, Diehl J. [Efficacy of caregiver support groups for dementia]. Nervenarzt. 2005 Mar;76(3):261-9. doi: 10.1007/s00115-004-1759-7. German. PMID 15300316
- [Background] Heinrich S, Laporte Uribe F, Roes M, Hoffmann W, Thyrian JR, Wolf-Ostermann K, Holle B. Knowledge management in dementia care networks: a qualitative analysis of successful information and support strategies for people with dementia living at home and their family caregivers. Public Health. 2016 Feb;131:40-8. doi: 10.1016/j.puhe.2015.10.021. Epub 2015 Dec 21. PMID 26718421
- [Background] ZQP. (2018). Ein Jahr nach letzter Pflegereform: Pflegende Angehörige sehen Informationsbedarf. Retrieved from https://www.presseportal.de/pm/80067/3876592?utm_source=digest&utm_medium=email&utm_campaign=push
- [Background] Gomez JF, Curcio CL, Alvarado B, Zunzunegui MV, Guralnik J. Validity and reliability of the Short Physical Performance Battery (SPPB): a pilot study on mobility in the Colombian Andes. Colomb Med (Cali). 2013 Sep 30;44(3):165-71. eCollection 2013 Jul. PMID 24892614
- [Background] Mendes MF, Tilbery CP, Balsimelli S, Moreira MA, Cruz AM. [Box and block test of manual dexterity in normal subjects and in patients with multiple sclerosis]. Arq Neuropsiquiatr. 2001 Dec;59(4):889-94. doi: 10.1590/s0004-282x2001000600010. Portuguese. PMID 11733833
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Spiegel R, Brunner C, Ermini-Funfschilling D, Monsch A, Notter M, Puxty J, Tremmel L. A new behavioral assessment scale for geriatric out- and in-patients: the NOSGER (Nurses' Observation Scale for Geriatric Patients). J Am Geriatr Soc. 1991 Apr;39(4):339-47. doi: 10.1111/j.1532-5415.1991.tb02897.x. PMID 2010583
- [Background] Bruce-Keller AJ, Brouillette RM, Tudor-Locke C, Foil HC, Gahan WP, Nye DM, Guillory L, Keller JN. Relationship between cognitive domains, physical performance, and gait in elderly and demented subjects. J Alzheimers Dis. 2012;30(4):899-908. doi: 10.3233/JAD-2012-120025. PMID 22466001
- [Background] Zank, S., Schacke, C., & Leipold, B. (2006). Berliner Inventar zur Angehörigenbelastung - Demenz (BIZA - D). Kurzbeschreibung und grundlegende Kennwerte. Retrieved from http://www.hf.uni-koeln.de/data/gerontologie/File/BIZA-D.pdf
- [Derived] Heinrich S, Cavazzini C, Holle B. DESKK Study - Development and testing of a dementia-specific respite care concept with a mobility and counselling programme: study protocol. BMJ Open. 2019 Jun 14;9(6):e025932. doi: 10.1136/bmjopen-2018-025932. PMID 31203237
- See also: Official Project Website — https://www.dzne.de/forschung/studien/projekte-der-versorgungsforschung/deskk/